CLINICAL TRIAL: NCT00148941
Title: Safety, Immunogenicity and Consistency of 3 Manufacturing Lots of DTaP-IPV Vaccine Versus Separate Injections of GSK Biologicals' DTaP + Aventis Pasteur's IPV Administered as Booster Doses to Healthy Children 4-6 Years, Each Co-administered With Merck's MMR Vaccine
Brief Title: Immune Response and Safety Comparison of 3 Lots of GSK Biologicals' DTaP-IPV Candidate Vaccine to DTaP + IPV Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 213503/048
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Tetanus; Acellular Pertussis; Diphtheria
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Tetanus Toxoid; Diphtheria-Tetanus-acellular Pertussis Vaccines; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Masking Description: The study was conducted in an open manner except for the consistency lots of SB213503 vaccine that were double-blinded.

ARMS (4):
- SB213503 lot 1 + M-M-R Group (Experimental): Subjects aged 4 to 6 years received a dose of lot 1 of SB213503 vaccine and a dose of M-M-R II vaccine.
  SB213503 was administered by deep intramuscular injection in the left deltoid. M-M-R II was co-administered as a subcutaneous injection in the upper right deltoid.
  Interventions: Biological: SB213503 lot 1; Biological: M-M-R II
- SB213503 lot 2 + M-M-R Group (Experimental): Subjects aged 4 to 6 years received a dose of lot 2 of SB213503 vaccine and a dose of M-M-R II vaccine.
  SB213503 was administered by deep intramuscular injection in the left deltoid. M-M-R II was co-administered as a subcutaneous injection in the upper right deltoid.
  Interventions: Biological: SB213503 lot 2; Biological: M-M-R II
- SB213503 lot 3 + M-M-R Group (Experimental): Subjects aged 4 to 6 years received a dose of lot 3 of SB213503 vaccine and a dose of M-M-R II vaccine.
  SB213503 was administered by deep intramuscular injection in the left deltoid. M-M-R II was co-administered as a subcutaneous injection in the upper right deltoid.
  Interventions: Biological: SB213503 lot 3; Biological: M-M-R II
- Infanrix + IPOL + M-M-R Group (Active Comparator): Subjects aged 4 to 6 years received a dose of Infanrix and a dose of IPOL vaccines separately and a dose of M-M-R II vaccine. Infanrix was administered by deep intramuscular injection in the upper left deltoid. IPOL was administered subcutaneously in the lower right deltoid. M-M-R II was co-administered as a subcutaneous injection in the upper right deltoid.
  Interventions: Biological: Infanrix; Biological: IPOL; Biological: M-M-R II

INTERVENTIONS:
Biological: SB213503 lot 1 — SB213503 lot 1 vaccine was administered as a single dose by intramuscular injection in the deltoid at Day 0.
  Other Names: GSK Biologicals combined diphteria, tetanus, acellular pertussis and inactivated poliovirus lot 1 vaccine
  Arms: SB213503 lot 1 + M-M-R Group
Biological: SB213503 lot 2 — SB213503 lot 2 vaccine was administered as a single dose by intramuscular injection in the deltoid at Day 0.
  Other Names: GSK Biologicals combined diphteria, tetanus, acellular pertussis and inactivated poliovirus lot 2 vaccine
  Arms: SB213503 lot 2 + M-M-R Group
Biological: SB213503 lot 3 — SB213503 lot 3 vaccine was administered as a single dose by intramuscular injection in the deltoid at Day 0.
  Other Names: GSK Biologicals combined diphteria, tetanus, acellular pertussis and inactivated poliovirus lot 3 vaccine
  Arms: SB213503 lot 3 + M-M-R Group
Biological: Infanrix — Infanrix vaccine was administered as a single dose by intramuscular injection in the deltoid at Day 0.
  Other Names: GSK Biologicals combined diphteria, tetanus, acellular pertussis vaccine
  Arms: Infanrix + IPOL + M-M-R Group
Biological: IPOL — IPOL vaccine was administered as a single dose by subcutaneous injection in the deltoid at Day 0.
  Other Names: Aventis Pasteur inactivated poliovirus vaccine
  Arms: Infanrix + IPOL + M-M-R Group
Biological: M-M-R II — M-M-R II vaccine was administered as a single dose by subcutaneous injection in the deltoid at Day 0.
  Other Names: Merck and Company licensed combined measles-mumps-rubella vaccine

SUMMARY:
The aims of this trial are to demonstrate the consistency of three manufacturing lots of GSK Biologicals' DTaP-IPV candidate vaccine in terms of immunogenicity and to evaluate the non-inferiority of GSK Biologicals' DTaP-IPV vaccine with respect to immunogenicity and safety compared to the control vaccines (separate injections of GSK Biologicals' DTaP vaccine [Infanrix] and Aventis Pasteur's IPV vaccine [IPOL]) when administered as a 5th dose of DTaP and a 4th dose of inactivated poliovirus vaccine in subjects 4 to 6 years of age. Vaccines will be co-administered with the second dose of M-M-RII, which is recommended at this age. Concomitant administration of a US-licensed influenza vaccine will be allowed according to seasonal availability of vaccine and at the discretion of the investigator.

DETAILED DESCRIPTION:
* Investigational groups: 3, each receive one of 3 lots of DTaP-IPV vaccine.
* Control: US-licensed DTaP (Infanrix) + US-licensed IPV (IPOL) vaccines administered in separate injections.
* Two study visits one month apart for a subset of subjects (Safety and Immunogenicity subset) with a blood draw at each visit. All other subjects will have one visit.
* A telephone contact 4-6 days after vaccination for all subjects, a telephone contact 31-38 days after vaccination for the Safety only subset and a telephone contact for all subjects during the extended safety follow-up phase (5 months following the active phase).

ELIGIBILITY:
Inclusion criteria:

* Male or female child between and including 4 and 6 years of age at the time of vaccination.
* Free of obvious health problems as established by medical history and brief medical evaluation before entering into the study.
* Received 4 doses of Infanrix and 3 doses of IPOL during the first 2 years of life.
* Vaccination against measles, mumps, and rubella in the second year of life.
* Subjects whom the investigator believed would comply with the requirements of the protocol.
* Written informed consent obtained before study entry from the parent(s) or guardian(s) of the subject.

Exclusion criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the administration of study vaccines, or planned use during the study period.
* History of previous or intercurrent diphtheria, tetanus, pertussis, polio, measles, mumps, or rubella disease, or of vaccination against these diseases given after the second year of life.
* Known exposure to diphtheria, tetanus, pertussis, or polio, prior to vaccination.
* Poliovirus vaccination with one or more doses of OPV vaccine.
* Administration or planned administration of a vaccine not foreseen by the study protocol within 30 days of study vaccination and ending at Day 30.
* Chronic administration or administration of immunosuppressants or other immune modifying drugs within six months prior to study vaccination or planned administration during the study period ending at Day 30.
* Administration of immunoglobulins and/or any blood products within three months prior to study vaccination or planned administration during the study period ending at Day 30.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection.
* History of seizures or progressive neurological disorder, including infantile spasms, uncontrolled epilepsy or progressive encephalopathy.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrollment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s), including allergic reactions to 2-phenoxyethanol, formaldehyde, neomycin, polymyxin B, streptomycin, gelatin, and/or latex.
* History of anaphylactic reaction to egg proteins or previous doses of the vaccine(s).
* Encephalopathy within 7 days of administration of previous dose of Infanrix.
* Fever ≥ 40.5°C or 104.9°F (rectal temperature) (39.5°C or 103.1°F, oral/axillary) within 48 hours of previous dose of Infanrix not due to another identifiable cause.
* Collapse or shock-like state (hypotonic-hyporesponsive episode) within 48 hours of previous dose of Infanrix.
* Persistent, severe, inconsolable screaming or crying lasting ≥ 3 hours which occurred within 48 hours of administration of previous dose of Infanrix.
* Thrombocytopenia following a previous dose of M-M-RII or its component vaccines.
* Inability to contact a parent/guardian of the subject by telephone.
* Blood dyscrasias (including current thrombocytopenia), leukemia, lymphomas or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Family history of congenital or hereditary immunodeficiency, unless the immune competence of the subject was demonstrated.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4209 (Actual)
Dates: Start 2005-01-06 (Actual); Primary Completion 2006-11-01 (Actual); Study Completion 2006-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (23):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Antioch, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fairfield, California
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Richmond, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, San Ramon, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Vacaville, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Mechanicsville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=368

REFERENCES:
- [Background] Black S, Friedland LR, Ensor K, Weston WM, Howe B, Klein NP. Diphtheria-tetanus-acellular pertussis and inactivated poliovirus vaccines given separately or combined for booster dosing at 4-6 years of age. Pediatr Infect Dis J. 2008 Apr;27(4):341-6. doi: 10.1097/INF.0b013e3181616180. PMID 18316985
- [Background] Weston WM, Klein NP. Kinrix: a new combination DTaP-IPV vaccine for children aged 4-6 years. Expert Rev Vaccines. 2008 Nov;7(9):1309-20. doi: 10.1586/14760584.7.9.1309. PMID 18980534
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 213503/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 213503/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 213503/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 213503/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 213503/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 213503/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 24 centers in the United States.
Pre-assignment Details: All 4209 subjects enrolled in the study, received the study vaccination and were included in the Total vaccination cohort (TVC).
Period: Overall Study
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Started | 1053 | 1051 | 1052 | 1053
Completed | 1035 | 1027 | 1032 | 1029
Not Completed | 18 | 24 | 20 | 24
Not completed — Lost to Follow-up | 17 | 24 | 18 | 22
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group | Total
Number analyzed (Participants) | 1053 | 1051 | 1052 | 1053 | 4209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.2 (0.38) | 4.2 (0.37) | 4.2 (0.37) | 4.2 (0.38) | 4.2 (0.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 526 | 515 | 533 | 513 | 2087
  Male | 527 | 536 | 519 | 540 | 2122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 65 | 74 | 77 | 77 | 293
  Race: White/Caucasian | 489 | 488 | 486 | 457 | 1920
  Race: Arabic/North African | 9 | 5 | 6 | 10 | 30
  Race: East/South East Asian | 83 | 95 | 75 | 103 | 356
  Race: South Asian | 45 | 51 | 55 | 50 | 201
  Race: American Hispanic | 208 | 201 | 188 | 194 | 791
  Race: Japanese | 3 | 5 | 3 | 4 | 15
  Race: Not specified | 151 | 132 | 162 | 158 | 603

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMCs) for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies in a Subset of Subjects
Description: GMCs were measured by Enzyme-Linked Immunosorbent assay (ELISA), expressed in international units per milliliter (IU/mL).
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: The anaylsis was performed on a subset of subjects (first 1340 enrolled subjects who agreed to participate in the subset) belonging to the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects who received study vaccines according to protocol and for whom immunogenicity data were available for the analyzed antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 284 | 283 | 284 | 261
IU/mL
  Anti-D: number analyzed (Participants) | 284 | 282 | 284 | 260
  Anti-D | 16.704 [15.198 to 18.360] | 18.658 [17.045 to 20.424] | 18.437 [16.771 to 20.269] | 18.112 [16.443 to 19.949]
  Anti-T | 9.693 [8.843 to 10.624] | 9.974 [9.120 to 10.908] | 11.300 [10.264 to 12.441] | 11.235 [10.275 to 12.284]
Statistical Analysis 1: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group; The lot-to-lot consistency of three manufacturing lots of SB213503 vaccine in terms of diphtheria toxoid (D) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Equivalence — Lot-to-lot consistency in terms of immunogenicity would be demonstrated if the lower and upper limits of the 95% confidence intervals (CIs) for the ratios of GMCs for each antigen (D, T, PT, FHA, PRN, and Poliovirus types 1, 2, and 3) and between each pair of the three lots of SB213503 vaccine were within the pre-defined clinical limits of [0.67; 1.5]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.970, 95% CI 2-sided [0.871 to 1.080]
Statistical Analysis 2: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Lot-to-lot consistency in terms of immunogenicity would be demonstrated if the lower and upper limits of the 95% CIs for the ratios of GMCs for each antigen (D, T, PT, FHA, PRN, and Poliovirus types 1, 2, and 3) and between each pair of the three lots of SB213503 vaccine were within the pre-defined clinical limits of [0.67; 1.5]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.961, 95% CI 2-sided [0.863 to 1.070]
Statistical Analysis 3: Comparison: SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.991, 95% CI 2-sided [0.890 to 1.103]
Statistical Analysis 4: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group; The lot-to-lot consistency of three manufacturing lots of SB213503 vaccine in terms of tetanus toxoid (T) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.975, 95% CI 2-sided [0.866 to 1.097]
Statistical Analysis 5: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.878, 95% CI 2-sided [0.780 to 0.988]
Statistical Analysis 6: Comparison: SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.901, 95% CI 2-sided [0.800 to 1.014]

2. Primary Outcome: Geometric Mean Concentrations (GMCs) for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibodies in a Subset of Subjects
Description: GMCs were measured by Enzyme-Linked Immunosorbent assay (ELISA), expressed in ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: The anaylsis was performed on a subset of subjects (first 1340 enrolled subjects who agreed to participate in the subset) belonging to the ATP cohort for immunogenicity, which included all evaluable subjects who received study vaccines according to protocol and for whom immunogenicity data were available for the analyzed antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 285 | 281 | 285 | 261
EL.U/mL
  Anti-PT: number analyzed (Participants) | 285 | 280 | 284 | 261
  Anti-PT | 66.9 [61.1 to 73.3] | 74.1 [66.6 to 82.4] | 71.4 [64.7 to 78.6] | 80.4 [72.4 to 89.1]
  Anti-FHA: number analyzed (Participants) | 285 | 280 | 285 | 261
  Anti-FHA | 809.1 [740.5 to 884.2] | 918.8 [840.0 to 1005.0] | 869.2 [795.2 to 950.2] | 939.7 [858.3 to 1028.8]
  Anti-PRN | 617.4 [549.2 to 694.0] | 584.7 [519.7 to 657.9] | 594.2 [526.6 to 670.4] | 593.8 [525.7 to 670.7]
Statistical Analysis 1: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group; The lot-to-lot consistency of three manufacturing lots of SB213503 vaccine in terms of pertussis toxoid (PT) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.938, 95% CI 2-sided [0.828 to 1.063]
Statistical Analysis 2: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.963, 95% CI 2-sided [0.850 to 1.091]
Statistical Analysis 3: Comparison: SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 1.026, 95% CI 2-sided [0.906 to 1.162]
Statistical Analysis 4: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group; The lot-to-lot consistency of three manufacturing lots of SB213503 vaccine in terms of filamentous haemagglutinin (FHA) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.874, 95% CI 2-sided [0.783 to 0.976]
Statistical Analysis 5: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 2, analysis 4]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.947, 95% CI 2-sided [0.849 to 1.057]
Statistical Analysis 6: Comparison: SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 2, analysis 4]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 1.084, 95% CI 2-sided [0.971 to 1.209]
Statistical Analysis 7: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group; The lot-to-lot consistency of three manufacturing lots of SB213503 vaccine in terms of pertactin (PRN) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 0.998, 95% CI 2-sided [0.867 to 1.148]
Statistical Analysis 8: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 2, analysis 7]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 1.043, 95% CI 2-sided [0.907 to 1.200]
Statistical Analysis 9: Comparison: SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 2, analysis 7]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance with more than 2 groups; GMC ratio = 1.045, 95% CI 2-sided [0.909 to 1.202]

3. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-poliovirus Types 1, 2 and 3 Antibodies in a Subset of Subjects
Description: GMTs were measured by Neutralization assay and expressed in titers.
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 276 | 274 | 276 | 252
Titers
  Anti-poliovirus 1: number analyzed (Participants) | 275 | 274 | 276 | 249
  Anti-poliovirus 1 | 2095.0 [1852.1 to 2369.8] | 2103.1 [1863.4 to 2373.5] | 2129.2 [1889.2 to 2399.7] | 1683.1 [1444.7 to 1960.9]
  Anti-poliovirus 2: number analyzed (Participants) | 276 | 273 | 269 | 252
  Anti-poliovirus 2 | 2345.4 [2104.8 to 2613.5] | 2132.9 [1888.0 to 2409.5] | 2326.6 [2074.5 to 2609.3] | 1802.0 [1566.3 to 2073.2]
  Anti-poliovirus 3: number analyzed (Participants) | 271 | 259 | 268 | 239
  Anti-poliovirus 3 | 3683.5 [3283.4 to 4132.3] | 3400.7 [3023.2 to 3825.4] | 3603.8 [3185.1 to 4077.5] | 3367.8 [2923.3 to 3879.8]
Statistical Analysis 1: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group; The lot-to-lot consistency of three manufacturing lots of SB213503 vaccine in terms of poliovirus type 1 geometric mean titers (GMTs) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Equivalence — Lot-to-lot consistency in terms of immunogenicity would be demonstrated if the lower and upper limits of the 95% CIs for the ratios of GMTs for each antigen (D, T, PT, FHA, PRN, and Poliovirus types 1, 2, and 3) and between each pair of the three lots of SB213503 vaccine were within the pre-defined clinical limits of [0.67; 1.5]; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 0.994, 95% CI 2-sided [0.836 to 1.181]
Statistical Analysis 2: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 0.987, 95% CI 2-sided [0.831 to 1.172]
Statistical Analysis 3: Comparison: SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 0.993, 95% CI 2-sided [0.836 to 1.180]
Statistical Analysis 4: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group; The lot-to-lot consistency of three manufacturing lots of SB213503 vaccine in terms of poliovirus type 2 geometric mean titers (GMTs) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 1.118, 95% CI 2-sided [0.951 to 1.314]
Statistical Analysis 5: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 3, analysis 4]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 1.006, 95% CI 2-sided [0.856 to 1.183]
Statistical Analysis 6: Comparison: SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 3, analysis 4]; Test type: Equivalence — Lot-to-lot consistency in terms of immunogenicity would be demonstrated if the lower and upper limits of the 95% CIs for the ratios of GMTs for each antigen (D, T, PT, FHA, PRN, and Poliovirus types 1, 2, and 3) and between each pair of the three lots of SB213503 vaccine were within the pre-defined clinical limits of [0.67; 1.5] for Anti-poliovirus type 2; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 0.900, 95% CI 2-sided [0.765 to 1.060]
Statistical Analysis 7: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group; The lot-to-lot consistency of three manufacturing lots of SB213503 vaccine in terms of poliovirus type 3 geometric mean titers (GMTs) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 1.112, 95% CI 2-sided [0.941 to 1.314]
Statistical Analysis 8: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 3, analysis 7]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 1.034, 95% CI 2-sided [0.876 to 1.220]
Statistical Analysis 9: Comparison: SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group; [analysis description as in outcome 3, analysis 7]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titer - pooled variance with more than 2 groups; GMT ratio = 0.930, 95% CI 2-sided [0.787 to 1.099]
Statistical Analysis 10: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Analysis of the non-inferiority of SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of anti-poliovirus type 1 (measured by the GMT ratio of Infanrix + IPOL + M-M-R Group over SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Non-Inferiority — The objectives were achieved if for D, T, PT, FHA and PRN: the upper limit of the two-sided standardized asymptotic 95% CI of the difference in booster response rates was less than or equal to the pre-defined clinical limit of 10% AND for poliovirus types 1, 2 and 3: the upper limit of the two-sided 95% confidence interval (CI) for the GMT ratio was less than or equal to the pre-defined clinical limit of 1.5; ANCOVA; ANCOVA model: adjustment for baseline titer - pooled variance; GMT ration = 0.792, 95% CI 2-sided [0.680 to 0.922]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis
Statistical Analysis 11: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Analysis of the non-inferiority of SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of anti-poliovirus type 2 (measured by the GMT ratio of Infanrix + IPOL + M-M-R Group over SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; ANCOVA; ANCOVA model: adjustment for baseline titer - pooled variance; GMT ratio = 0.802, 95% CI 2-sided [0.696 to 0.925]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis
Statistical Analysis 12: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Analysis of the non-inferiority of SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of anti-poliovirus type 3 (measured by the GMT ratio of Infanrix + IPOL + M-M-R Group over SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; ANCOVA; ANCOVA model: adjustment for baseline titer - pooled variance; GMT ratio = 0.938, 95% CI 2-sided [0.811 to 1.085]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis

4. Primary Outcome: Number of Subjects With Booster Response Against Diphtheria Toxoid (D) and Tetanus Toxoid (T) Antigens in a Subset of Subjects
Description: Vaccine response defined as: For initially seronegative subjects [pre-booster antibody concentration below (<) cut-off of 0.1 international units per milliliter (IU/mL)] with an increase of at least four times the cut-off one month after vaccination [post-booster antibody concentration greater than or equal to (≥) 0.4 IU/mL]. For initially seropositive subjects (pre-booster antibody concentration ≥ 0.1 IU/mL) with an increase of at least four times the pre-booster antibody concentration one month after vaccination.
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: The analysis was performed on a subset of subjects (first 1340 enrolled subjects who agreed to participate in the subset) belonging to the ATP cohort for immunogenicity, which included all evaluable subjects who received study vaccines according to protocol and for whom immunogenicity data were available for the analyzed antigen.
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 280 | 283 | 282 | 261
Participants
  Anti-D, Total: number analyzed (Participants) | 280 | 282 | 282 | 260
  Anti-D, Total | 279 | 280 | 281 | 260
  Anti-T, Total: number analyzed (Participants) | 279 | 283 | 282 | 261
  Anti-T, Total | 266 | 273 | 277 | 245
Statistical Analysis 1: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Analysis of the non-inferiority of SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of diphtheria toxoid (D) booster responses (i.e measured by the difference in percentage of subjects with a booster response between the Infanrix + IPOL + M-M-R Group and (minus) the SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; Difference between groups = 0.47, 95% CI 2-sided [-0.98 to 1.21]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis
Statistical Analysis 2: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Analysis of the non-inferiority of SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of tetanus toxoid (T) booster responses (measured by the difference in percentage of subjects with a booster response between the Infanrix + IPOL + M-M-R Group and (minus) the SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; Difference between groups = -2.81, 95% CI 2-sided [-6.55 to -0.09]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis

5. Primary Outcome: Number of Subjects With Booster Response Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) Antigens in a Subset of Subjects
Description: Vaccine response defined as: For initially seronegative subjects [pre-booster antibody concentration below (<) cut-off of 5 EL.U/mL] with an increase of at least four times the cut-off one month after vaccination (post-booster antibody concentration ≥ 20 EL.U/mL). For initially seropositive subjects with pre-booster antibody concentration ≥ 5 EL.U/mL and < 20 EL.U/mL with an increase of at least 4 times the pre-booster antibody concentration one month after vaccination. For initially seropositive subjects with pre-booster antibody concentration ≥ 20 EL.U/mL with an increase of at least 2 times the pre-booster antibody concentration one month after vaccination.
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 281 | 281 | 284 | 261
Participants
  Anti-PT, Total: number analyzed (Participants) | 272 | 273 | 277 | 256
  Anti-PT, Total | 251 | 250 | 257 | 237
  Anti-FHA, Total: number analyzed (Participants) | 281 | 280 | 283 | 261
  Anti-FHA, Total | 265 | 272 | 268 | 251
  Anti-PRN, Total: number analyzed (Participants) | 280 | 281 | 284 | 261
  Anti-PRN, Total | 270 | 277 | 279 | 253
Statistical Analysis 1: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Analysis of the non-inferiority of SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of pertussis toxoid (PT) booster responses (measured by the difference in percentage of subjects with a booster response between the Infanrix + IPOL + M-M-R Group and (minus) the SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; Difference between groups = 0.36, 95% CI 2-sided [-3.83 to 3.71]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis
Statistical Analysis 2: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Analysis of the non-inferiority of SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of filamentous haemagglutinin (FHA) booster responses (measured by the difference in percentage of subjects with a booster response between the Infanrix + IPOL + M-M-R Group and (minus) the SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; Difference between groups = 0.79, 95% CI 2-sided [-2.50 to 3.21]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis
Statistical Analysis 3: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Analysis of the non-inferiority of SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of pertactin (PRN) booster responses (measured by the difference in percentage of subjects with a booster response between the Infanrix + IPOL + M-M-R Group and (minus) the SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups) in a subset of subjects one month after vaccination when co-administered with M-M-R II; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; Difference between groups = -0.82, 95% CI 2-sided [-3.79 to 1.14]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis

6. Primary Outcome: Number of Subjects With Circumferential Swelling at the Injection Site
Description: Swelling (at the SB213503 & Infanrix injection sites) was categorized as an increase of > or ≤ 30 mm in mid upper arm circumference compared to baseline measurement or with an increase in mid upper arm missing; extent of swelling > or ≤ 50 % of upper arm length, or diameter of injection site missing.
Time Frame: Within 4 days (Day 0-3) after vaccination
Population: The analysis was performed on the Total vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1053 | 1051 | 1052 | 1053
Participants
  Circumference increase>30mm;swelling>50% of length | 5 | 10 | 5 | 11
  Circumference increase>30mm;swelling≤50% of length | 10 | 20 | 23 | 22
  Circumference increase>30mm;diameter missing | 2 | 0 | 1 | 1
  Circumference increase≤30mm;swelling>50% of length | 9 | 10 | 12 | 12
  Circumference increase≤30mm;swelling≤50% of length | 62 | 42 | 52 | 54
  Circumference increase≤30mm;diameter missing | 0 | 0 | 0 | 0
  Increase in mid upper arm;swelling>50% of length | 0 | 0 | 0 | 0
  Increase in mid upper arm;swelling≤50% of length | 0 | 2 | 0 | 0
  Increase in mid upper arm;diameter missing | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: SB213503 Lot 1 + M-M-R Group vs SB213503 Lot 2 + M-M-R Group vs SB213503 Lot 3 + M-M-R Group vs Infanrix + IPOL + M-M-R Group; Non-inferiority of the SB213503 vaccine compared to Infanrix + IPOL administered separately in terms of the incidence of increased circumferential swelling at the SB213503 and Infanrix injection site, defined as an injection site swelling diameter that involves > 50% of the length of the upper arm that also is associated with a > 30 mm increase of the mid-upper arm circumference compared to the baseline measurement; Test type: Non-Inferiority — Non-inferiority objective was considered demonstrated, when the upper limit of the 95% CI for the difference between groups (SB213503 + M-M-R Group = pooled lot 1, 2 & 3 groups minus Infanrix + IPOL + M-M-R Group) in percentage of subjects reporting increased circumferential swelling was equal or less than 2%; Difference in percentage = -0.41, 95% CI 2-sided [-1.26 to 0.16]; SB213503 lot 1, SB213503 lot 2, and SB213503 lot 3 Arms/Groups were pooled for statistical analysis

7. Secondary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Antigens in a Subset of Subjects
Description: A seroprotected subject is defined as a vaccinated subject with anti-D and anti-T antibody concentration greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 284 | 283 | 284 | 261
Participants
  Anti-D: number analyzed (Participants) | 284 | 282 | 284 | 260
  Anti-D | 284 | 282 | 284 | 260
  Anti-T | 284 | 283 | 284 | 261

8. Secondary Outcome: Number of Seroprotected Subjects Against Poliovirus Types 1, 2 and 3 Antigens in a Subset of Subjects
Description: A seroprotected subject is defined as a vaccinated subject with anti-poliovirus types 1, 2 and 3 antibody titers greater than or equal to 1:8.
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 276 | 274 | 276 | 252
Participants
  Anti-poliovirus type 1: number analyzed (Participants) | 275 | 274 | 276 | 249
  Anti-poliovirus type 1 | 275 | 274 | 275 | 249
  Anti-poliovirus type 2: number analyzed (Participants) | 276 | 273 | 269 | 252
  Anti-poliovirus type 2 | 276 | 273 | 269 | 252
  Anti-poliovirus type 3: number analyzed (Participants) | 271 | 259 | 268 | 239
  Anti-poliovirus type 3 | 271 | 259 | 268 | 239

9. Secondary Outcome: Number of Seropositive Subjects Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) Antigens in a Subset of Subjects
Description: A seropositive subject was defined as a vaccinated subject with anti-PT, anti-FHA and anti-PRN antibody concentrations greater than or equal to (≥) 5 ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 285 | 281 | 285 | 261
Participants
  Anti-PT: number analyzed (Participants) | 285 | 280 | 284 | 261
  Anti-PT | 285 | 279 | 283 | 261
  Anti-FHA: number analyzed (Participants) | 285 | 280 | 285 | 261
  Anti-FHA | 285 | 280 | 285 | 261
  Anti-PRN | 285 | 281 | 285 | 261

10. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations Greater Than or Equal to (≥) 1 IU/mL
Description: The number of subjects with anti-D and anti-T antibody concentrations greater than or equal to (≥) 1 IU/mL is reported.
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 284 | 283 | 284 | 261
Participants
  Anti-D: number analyzed (Participants) | 284 | 282 | 284 | 260
  Anti-D | 284 | 282 | 284 | 260
  Anti-T | 281 | 282 | 281 | 261

11. Secondary Outcome: Number of Subjects With Booster Response for Poliovirus Types 1, 2 and 3 Antigens in a Subset of Subjects
Description: Vaccine response defined as: For initially seronegative subjects (pre-booster antibody titer below cut-off of 1:8), an antibody titer ≥ 1:32 at one month after vaccination. For initially seropositive subjects (pre-booster antibody titer ≥1:8), an increase at least four times the pre-booster antibody titer at one month after vaccination.
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 274 | 268 | 273 | 252
Participants
  Anti-poliovirus type 1, Total: number analyzed (Participants) | 270 | 266 | 273 | 249
  Anti-poliovirus type 1, Total | 264 | 257 | 264 | 231
  Anti-poliovirus type 2, Total: number analyzed (Participants) | 274 | 268 | 265 | 252
  Anti-poliovirus type 2, Total | 271 | 252 | 258 | 234
  Anti-poliovirus type 3, Total: number analyzed (Participants) | 269 | 255 | 263 | 237
  Anti-poliovirus type 3, Total | 259 | 245 | 256 | 220

12. Secondary Outcome: Geometric Mean Titers (GMTs) for Serum Haemagglutination-inhibition (HI) Anti-H1N1, Anti-H3N2 and Anti-B Antibodies in a Subset of Subjects
Description: GMTs were measured by hemagglutination inhibition assay and expressed in titers.
Time Frame: At Day 0 (i.e. before vaccination) and at Month 1 (i.e. one month after vaccination)
Population: The analysis was performed on a subset of subjects (first 1340 enrolled subjects who agreed to participate in the subset) belonging to the ATP cohort for immunogenicity, which included all evaluable subjects who received concomitant influenza vaccine and for whom immunogenicity data were available for the analyzed antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1 | 4 | 2 | 2
Titers
  Anti-H1N1, Day 0: number analyzed (Participants) | 1 | 3 | 2 | 2
  Anti-H1N1, Day 0 | 5.0 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable) because number of subjects with concentrations within the specified range = 0. | 20.0 [0.1 to 7789.1] | 20.0 [0.0 to 893160000] | 56.6 [0.0 to NA] — NA=1.38*10^15 in this case
  Anti-H1N1, Month 1 | 57.0 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable) because number of subjects with concentrations within the specified range = 0. | 134.5 [25.7 to 703.7] | 20.0 [0.0 to 133653.0] | 226.3 [0.0 to 826100000000]
  Anti-H3N2, Day 0: number analyzed (Participants) | 1 | 3 | 2 | 2
  Anti-H3N2, Day 0 | 1280.0 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable) because number of subjects with concentrations within the specified range = 0. | 80.0 [0.2 to 31156.2] | 80.0 [0.0 to NA] — NA=1.595*10^17 in this case | 134.5 [14.8 to 1225.1]
  Anti-H3N2, Month 1 | 1280.0 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable) because number of subjects with concentrations within the specified range = 0. | 493.6 [61.6 to 3958.1] | 113.1 [0.0 to NA] — NA=2.76*10^15 in this case | 538.1 [0.7 to 397480.8]
  Anti-B, Day 0: number analyzed (Participants) | 1 | 3 | 2 | 2
  Anti-B, Day 0 | 160.0 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable) because number of subjects with concentrations within the specified range = 0. | 10.0 [0.5 to 197.3] | 7.1 [0.1 to 578.0] | 10.0 [0.0 to 66826.5]
  Anti-B, Month 1 | 1810.0 [NA to NA] — The lower limit (LL) and upper limit (UL) of the 95% confidence interval could not be determined in this group (not applicable) because number of subjects with concentrations within the specified range = 0. | 95.1 [9.8 to 924.4] | 28.3 [0.3 to 2312.2] | 226.3 [0.0 to 826100000000]

13. Secondary Outcome: Number of Seroconverted Subjects Against Influenza Virus Strains H1N1, H3N2, and B in a Subset of Subjects
Description: Seroconversion was defined as a post-vaccination haemagglutination-inhibition (HI) titer of ≥ 1:40 in an initially HI antibody seronegative subject (pre-vaccination HI titer < 1:10), or a ≥ 4 fold rise in HI titer in an initially HI antibody seropositive subject (pre-vaccination HI titer ≥ 1:10) The 3 flu strains assessed were H1N1, H3N2, and B.
Time Frame: At Month 1 (i.e. one month after vaccination)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1 | 3 | 2 | 2
Participants
  Anti-H1N1 | 1 | 2 | 0 | 1
  Anti-H3N2 | 0 | 2 | 0 | 1
  Anti-B | 1 | 3 | 1 | 2

14. Secondary Outcome: Number of Seroprotected Subjects Against Influenza Virus Strains H1N1, H3N2, and B in a Subset of Subjects
Description: A seroprotected subject is defined as a vaccinated subject with anti-H1N1, anti-H3N2, and anti-B antibody titers greater than or equal to (≥) 1:40.
Time Frame: At Day 0 (i.e. before vaccination) and at Month 1 (i.e. one month after vaccination)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1 | 4 | 2 | 2
Participants
  Anti-H1N1, Day 0: number analyzed (Participants) | 1 | 3 | 2 | 2
  Anti-H1N1, Day 0 | 0 | 1 | 1 | 1
  Anti-H1N1, Month 1 | 1 | 4 | 1 | 2
  Anti-H3N2, Day 0: number analyzed (Participants) | 1 | 3 | 2 | 2
  Anti-H3N2, Day 0 | 1 | 2 | 1 | 2
  Anti-H3N2, Month 1 | 1 | 4 | 1 | 2
  Anti-B, Day 0: number analyzed (Participants) | 1 | 3 | 2 | 2
  Anti-B, Day 0 | 1 | 1 | 0 | 0
  Anti-B, Month 1 | 1 | 3 | 1 | 2

15. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness, and swelling (at the SB213503 & Infanrix vaccination sites). Any = any symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activities. Grade 3 redness/swelling = redness/swelling spreading up to or beyond 50 mm diameter.
Time Frame: During the 4-day (Day 0-3) post-vaccination period
Population: The anaylsis was performed on the Total vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented and with symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1046 | 1039 | 1043 | 1043
Participants
  Pain, Any | 620 | 582 | 642 | 601
  Pain, Grade 3 | 19 | 17 | 13 | 7
  Redness, Any | 391 | 399 | 412 | 423
  Redness, Grade 3 | 187 | 186 | 194 | 213
  Swelling, Any | 295 | 266 | 291 | 296
  Swelling, Grade 3 | 111 | 95 | 118 | 122

16. Secondary Outcome: Number of Subjects With Any and Grade 3 Increase in the Mid-upper Arm Circumference at the Injection Site
Description: Assessed specific symptom was increase in mid upper arm circumference (at the SB213503 & Infanrix injection sites). Any = any symptom regardless of intensity grade. Grade 3 increase in mid upper arm circumference = mid upper arm circumference greater than 30 mm.
Time Frame: During the 4-day (Day 0-3) post-vaccination period
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1046 | 1039 | 1043 | 1043
Participants
  Increase in mid-upper arm circumference, Any | 368 | 374 | 393 | 397
  Increase in mid-upper arm circumference, Grade 3 | 16 | 29 | 29 | 33

17. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever (orally) [≥ 37.5 degrees Celsius (°C)] and loss of appetite. Any = any solicited general symptom irrespective of intensity grade or relationship to vaccination. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 loss of appetite = not eating at all. Related = considered by the investigator to be related to the vaccine. Grade 3 fever = fever >39°C.
Time Frame: During the 4-day (Day 0-3) post-vaccination period
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1044 | 1037 | 1040 | 1036
Participants
  Drowsiness, Any | 194 | 216 | 185 | 181
  Drowsiness, Grade 3 | 9 | 10 | 7 | 8
  Drowsiness, Related | 153 | 166 | 148 | 141
  Fever (orally), ≥ 37.5 °C | 167 | 154 | 166 | 147
  Fever (orally), > 39.0 °C | 9 | 8 | 16 | 11
  Fever (orally), Related | 154 | 136 | 143 | 128
  Loss of appetite, Any | 162 | 160 | 162 | 166
  Loss of appetite, Grade 3 | 11 | 6 | 7 | 6
  Loss of appetite, Related | 127 | 117 | 130 | 125

18. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms Specific to M-M-R II Vaccination
Description: Solicited general symptoms specific to M-M-R II vaccination were fever [≥ 37.5 degrees Celsius (°C)], rash/exanthem, parotid/salivary gland swelling, and suspected signs of meningism including febrile convulsions . Any = any symptom regardless of intensity grade. Grade 3 = symptom that prevented normal everyday activity. Related = considered by the investigator to be related to the vaccine. Grade 3 fever = fever >39°C.
Time Frame: During the 15-day (Day 0-14) post-vaccination period
Population: The analysis was performed on the Total vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented and with symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1044 | 1037 | 1040 | 1036
Participants
  Rash site, Any | 34 | 44 | 21 | 36
  Non-administration site rash, Measles/Rubella-like | 5 | 4 | 4 | 6
  Non-administration site rash, Grade 3 | 0 | 0 | 0 | 0
  Non-administration site rash, Related | 5 | 6 | 4 | 4
  Parotitis, Any | 1 | 3 | 2 | 3
  Suspected signs of meningism, Any | 7 | 5 | 4 | 5
  Fever (orally), ≥ 37.5°C | 213 | 215 | 218 | 208
  Fever (orally), > 39.0°C | 22 | 25 | 36 | 23
  Fever (orally), Related | 169 | 155 | 159 | 140

19. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Days 0-30) post-vaccination period
Population: The anaylsis was performed on the Total vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1053 | 1051 | 1052 | 1053
Participants | 321 | 317 | 326 | 307

20. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) that were assessed included medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: During the entire study period (from Day 0 through 6 months [minimum 182 days post-vaccination])
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1053 | 1051 | 1052 | 1053
Participants | 4 | 7 | 1 | 4

21. Secondary Outcome: Number of Subjects With Onset of Chronic Illness(es) and AE(s) Leading to Emergency Room (ER) or to Physician Office Visits
Description: Among assessed chronic illness(es) were: autoimmune disorders, asthma, type I diabetes, and allergies. AEs leading to emergency room (ER) visits or to physician office visits that were not related to well-child care, vaccination, injury or common acute illnesses such as upper respiratory tract infection, otitis media, pharyngitis, and gastroenteritis.
Time Frame: During the extended safety follow-up phase (i.e. 5 months following the active phase [from Day 31 up to minimum 182 days post-vaccination])
Population: The analysis was performed on the Extended Safety Follow Up (ESFU) cohort, which included all vaccinated subjects who had a follow-up contact during the ESFU period/who reported an unsolicited AE as specified in the protocol/onset of a chronic illness/SAE beyond Day 30, after the last vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
Number analyzed (Participants) | 1028 | 1019 | 1024 | 1022
Participants
  Chronic illness | 6 | 6 | 4 | 5
  Emergency room visit | 7 | 7 | 10 | 8
  Physician's office visit | 20 | 22 | 22 | 19

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Days 0-3) post-vaccination period; MMR II specific solicited symptoms: during the 15-day (Days 0-14) post-vaccination period; Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period; SAEs: during the entire study period (from Day 0 through 6 months [minimum 182 days post-vaccination]).
Arm/Group | SB213503 Lot 1 + M-M-R Group | SB213503 Lot 2 + M-M-R Group | SB213503 Lot 3 + M-M-R Group | Infanrix + IPOL + M-M-R Group
All-Cause Mortality (participants affected / at risk) | 0/1053 | 0/1051 | 0/1052 | 0/1053
Serious Adverse Events (participants affected / at risk) | 4/1053 | 7/1051 | 1/1052 | 4/1053
Other Adverse Events (participants affected / at risk) | 797/1053 | 783/1051 | 814/1052 | 804/1053
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB213503 Lot 1 + M-M-R Group (N=1053) | SB213503 Lot 2 + M-M-R Group (N=1051) | SB213503 Lot 3 + M-M-R Group (N=1052) | Infanrix + IPOL + M-M-R Group (N=1053)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia necrotizing (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB213503 Lot 1 + M-M-R Group (N=1053) | SB213503 Lot 2 + M-M-R Group (N=1051) | SB213503 Lot 3 + M-M-R Group (N=1052) | Infanrix + IPOL + M-M-R Group (N=1053)
Decreased appetite (Metabolism and nutrition disorders) | 162 (162) | 160 (160) | 162 (162) | 166 (166)
Erythema (Skin and subcutaneous tissue disorders) | 391 (392) | 400 (400) | 412 (412) | 424 (424)
Pain (General disorders) | 620 (622) | 583 (584) | 642 (642) | 601 (604)
Pyrexia (General disorders) | 227 (229) | 228 (232) | 234 (241) | 233 (236)
Somnolence (Nervous system disorders) | 194 (194) | 217 (217) | 185 (185) | 181 (181)
Swelling (General disorders) | 295 (295) | 266 (266) | 292 (292) | 298 (298)
Upper respiratory tract infection (Infections and infestations) | 54 (56) | 57 (59) | 71 (71) | 60 (63)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.